CLINICAL TRIAL: NCT00001332
Title: Phase I Study of Continuous Hyperthermic Peritoneal Perfusion (CHPP) With Escalating Dose I.P. Platinum for Gastrointestinal Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930048; 93-C-0048
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Peritoneal Neoplasms; Stomach Neoplasms
Keywords: Cancer Treatment; Chemotherapy; Regional Therapy; Surgery
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms | interventions — Cisplatin

INTERVENTIONS:
Procedure: CHPP with cisplatin

SUMMARY:
Patients with gastric adenocarcinoma are most frequently diagnosed at an advanced stage. The disease has a marked propensity for loco-regional spread and will be the sole or major site of disease in up to 80% of patients. Various attempts at controlling loco-regional disease have not been successful. The selective lethal effect of supranormal temperatures on neoplastic cells and the additive or synergistic effect of combining chemotherapy has been well established in laboratory models and has provided the rationale for numerous clinical trials using hyperthermic isolated limb perfusion for advanced extremity melanoma or sarcoma. This Phase I study will evaluate the safety of escalating temperatures of continuous hyperthermic peritoneal perfusion (CHPP) with escalating doses of intraperitoneal Cisplatin (CDDP) in the treatment of patients with advanced peritoneal adenocarcinoma of gastrointestinal origin.

DETAILED DESCRIPTION:
Patients with gastric adenocarcinoma are most frequently diagnosed at an advanced stage. The disease has a marked propensity for loco-regional spread and will be the sole or major site of disease in up to 80% of patients. Various attempts at controlling loco-regional disease have not been successful. The selective lethal effect of supranormal temperatures on neoplastic cells and the additive or synergistic effect of combining chemotherapy has been well established in laboratory models and has provided the rationale for numerous clinical trials using hyperthermic isolated limb perfusion for advanced extremity melanoma or sarcoma. This Phase I study will evaluate the safety of escalating temperatures of continuous hyperthermic peritoneal perfusion (CHPP) with escalating doses of intraperitoneal Cisplatin (CDDP) in the treatment of patients with advanced peritoneal adenocarcinoma of gastrointestinal origin.

ELIGIBILITY:
Patients age greater than or equal to 18 years.

Patients with histologically proven gastrointestinal adenocarcinoma, mesothelioma, or sarcoma. By standard staging studies there must be evidence of advanced or metastatic intraabdominal disease. Patients with minimal extraabdominal metastatic disease and who have symptoms exclusively referable to advanced intraabdominal malignancy will be considered for the study. Specifically, patients with gastric cancer and bulky N-2 lymph node involvement or patients with other primaries and who have malignant ascites or peritoneal seeding would be considered optimal candidates. If all gross peritoneal disease is resected (i.e., gross omental implants removed by gastrectomy), patients are still eligible for treatment.

Patients must have recovered from any toxicity from all prior chemotherapy, immunotherapy, or radiotherapy (30 days).

Patients must not have any significant systemic illness (e.g., infection, cardiovascular, or pulmonary) which would preclude them from being an operative candidate.

patients must have a life expectancy of at least 8 weeks.

Performance status should be ECOG level 0, 1, or 2.

Patients must have adequate renal function (i.e., serum creatinine less than or equal to 2.0 or creatinine clearance of greater than or equal to 45 ml/min).

Patients must be HIV negative.

Women of child bearing age must not be pregnant or breast feeding.

Patients with prior CDDP will be eligible if there is no evidence of existing irreversible CDDP toxicity. Patients suspected of having chronic CDDP toxicity will be further evaluated as clinically indicated.

Patients may have mild elevations (less than 2.0 times normal) in liver function test if the abnormalities are consistent with advanced intra-abdominal cancer.

Abnormalities (greater than 1 sec over normal) in PT or PTT or severe thrombocytopenia (less than 75 K) will render patients ineligible.

A low Hgb secondary to chronic tumor-related, blood loss is acceptable if the patient is willing and able to have transfusion.

Patients will be ineligible if the WBC is less than 3,000.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1992-12; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wisbeck WM, Becher EM, Russell AH. Adenocarcinoma of the stomach: autopsy observations with therapeutic implications for the radiation oncologist. Radiother Oncol. 1986 Sep;7(1):13-8. doi: 10.1016/s0167-8140(86)80120-7. PMID 3775075
- [Background] Eggermont AM, Sugarbaker PH. Efficacy of intracavitary administration of cyclophosphamide, interleukin-2 and lymphokine activated killer cells against established intraperitoneal tumor. Acta Med Austriaca. 1989;16(3-4):47-50. PMID 2609913
- [Background] Knusli C, Ruff P, Laffer U, Stoll HR, Obrist R, Weber W, Obrecht JP. Intraperitoneal chemotherapy in peritoneal malignancy: impact of intensive system care on practicability. Acta Med Austriaca. 1989;16(3-4):70-3. PMID 2692376